CLINICAL TRIAL: NCT05080088
Title: A Pilot Study: Retrospective Evaluation of 3 Colonic Adenoma Detection Strategies During a Colonoscopy: Endoscopy Cap Associated With the Artificial Intelligence GI GENIUS ™ System, the Artificial Intelligence GI GENIUS ™ Alone and Colonoscopy Alone
Brief Title: Retrospective Evaluation of 3 Colonic Adenoma Detection Strategies
Acronym: COLODETECT
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Principal Investigator, Clément Delliot, medical student, Centre Hospitalier Universitaire de Nīmes
Other Study IDs: 21.06.06
Record Dates: First submitted 2021-10-02; First posted 2021-10-15 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Adenoma Colon; Colorectal Cancer; Colorectal Polyp; Colonic Adenocarcinoma
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Colonoscopy Only Group
- Artificial intelligence GI GENIUS ™ only Group
- Endoscopic Cap and Artificial Intelligence GI GENIUS ™ Group

SUMMARY:
Retrospective study, single blind (patient), allowing a posteriori clinical data collection of 90 patients during their passage to the ambulatory endoscopy circuit, to consider 3 groups and thus to deduce a colonic adenoma detection rate for each arm :

* Colonoscopy Only Group
* Artificial intelligence only group (IA GI GENIUS ™ alone)
* Endoscopic Cap and Artificial Intelligence Group (endoscopy cap associated with the GI GENIUS ™ IA System)

ELIGIBILITY:
Inclusion Criteria :

* 18 years < Patient < 85 years
* Need to perform a primary and / or secondary screening colonoscopy for colorectal cancer
* Patients candidates for outpatient care

Exclusion Criteria :

* History of inflammatory digestive tract disease
* Failed previous colonoscopy
* Known familial polyposis
* Biopsy / polypectomy contraindication (coagulation disorder, treatment with CLOPIDOGREL / Anticoagulant)

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients are recruited during a pre-colonoscopy consultation, carried out by the gastroenterologist in current practice
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2021-04-06 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-08 (Actual)

PRIMARY OUTCOMES:
Colonic Adenomas Detection Rate according to the use of the Combine Techniques GENIUS software - Cap or Only GENIUS software | 4 months
  number of colonoscopies with the discovery of at least 1 colonic adenoma out of the total number of colonoscopies according to the use of colonoscopy alone / artificial intelligence alone / artificial intelligence combined with the endoscopic cap.

SECONDARY OUTCOMES:
Adenomas Rate according to their morphology | 4 months
  according to Paris classification
Adenomas Rate according to their size | 4 months
  < 0,5mm / 0-5-10mm / > 10mm
Adenomas Rate according to their histology | 4 months
  according to Vienne classification
Caecal Intubation Rate | 4 months
  Complete colonocopy rate
Withdrawal time | 4 months
Adverse effects | 4 months
  Haemorrhages, Perforation

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Nîmes, Nîmes, Gard, France

REFERENCES:
- [Derived] Caillo L, Delliot C, Chevallier T, Bourgaux JF, Prost A, Brunaud-Gagniard B, Phoutthasang V, Clerc C, Borderie T, Daniel J, Pouderoux P, Debourdeau A. COLODETECT 1: comparative evaluation of endocuff with computer-aided detection versus computer-aided detection alone versus standard colonoscopy for enhancing adenoma detection rates during screening colonoscopy-a pilot study. Therap Adv Gastroenterol. 2024 Oct 27;17:17562848241290433. doi: 10.1177/17562848241290433. eCollection 2024. PMID 39493261